CLINICAL TRIAL: NCT05197010
Title: Clinical Efficacy of IoMT-based Exercise Program for the Elderly With Chronic Musculoskeletal Disorders
Brief Title: Clinical Efficacy of IoMT-based Exercise Program for the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-04-004
Record Dates: First submitted 2021-12-08; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Lower Back Pain; Knee Osteoarthritis
MeSH Terms: conditions — Low Back Pain; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-blinded, two-armed randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator responsible for randomization was independent from the assessors, assuring blindness to treatment allocation and randomization procedures. The blinded assessor performed the baseline and post-treatment assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based exercise program (Experimental): The subjects will receive 6 weeks of the home exercise program via a smartphone application. The home exercise program sets the exercise intensity to 3 levels (low, medium, and high) according to the disease and consists of 2 stretches, 3 strengthening and/or functional exercises, and a cool-down exercise. The exercise group applies a daily home exercise program (30min/day, 7days/week for 6 weeks).
  Interventions: Other: Home based exercise program via a smartphone application
- Exercise brochure (No Intervention): This group will be offered a brochure including number of exercises for back or knee.

INTERVENTIONS:
Other: Home based exercise program via a smartphone application — Daily home based exercise program (30min/day, 7days/week for 6 weeks).
  Arms: Home-based exercise program

SUMMARY:
The purpose of this study is to evaluate the efficacy of Internet of Medical Things (IoMT) based home exercise programs for the elderly with degenerative knee arthritis or chronic low back pain.

DETAILED DESCRIPTION:
This study presents the protocol of a prospective, single-center, single-blinded, two-armed randomized controlled trial.

The investigators plan to recruit patients over 65 years of age with degenerative knee arthritis or chronic low back pain. Patients will be randomly divided into two groups with 1:1 allocation.

The intervention group will receive 6 weeks of the IoT-based home exercise program. The IoMT-based home exercise program is implemented to the patients via a smartphone application. The home exercise program sets the exercise intensity to 3 levels (low, medium, and high) according to the disease and consists of 2 stretches, 3 strengthening and/or functional exercises, and a cool-down exercise (Figure 1). The exercise group applies a daily home exercise program (30min/day, 7days/week for 6 weeks).

The activity detector records the amount of activity and the speed of movement within the home. The door sensor detects the enter and exit and records the number of outings. The pillbox notifies subjects to take the medication time. The smart-care phone provides emergency call and guardian connection services. The body composition analyzer measures body mass index, fat, and muscle mass.

The primary outcome in patients with degenerative knee arthritis is Western Ontario and McMaster Universities Osteoarthritis. And the primary outcome in patients with chronic low back pain is Oswestry Disability Index. The secondary outcomes are numeric rating scale for pain, 36-Item Short-Form Health Survey, Geriatric Depression Scale, Timed-Up and Go test, and 30s chair sit and stand.

The investigators evaluate primary and secondary outcomes before and after the home exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain for more than 3months, Kellgren-Lawrence grade 2 or higher
* Low back pain for more than 3months
* A person who underdtands the exercise program
* Numeric rating scale of 4 or higher

Exclusion Criteria:

* History of knee surgery
* Systemic inflammatary disease
* History of polyneuropathy
* History of stroke
* Severe heart failure
* Chronic obstructive pulmonary disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis | baseline
  Knee osteoarthritis functional index (Range: 0-96)
Western Ontario and McMaster Universities Osteoarthritis | after 6weeks
  Knee osteoarthritis functional index (Range: 0-96)
Oswestry Disability Index | baseline
  Low back pain functional index (Range: 0-100)
Oswestry Disability Index | after 6weeks
  Low back pain functional index (Range: 0-100)

SECONDARY OUTCOMES:
Numeric rating scale | baseline
  Pain score, The higher score means the worse pain (Range: 0-10)
Numeric rating scale | after 6weeks
  Pain score, The higher score means the worse pain (Range: 0-10)
36-Item Short-Form Health Survey | baseline
  Qualify of life, The higher score means the better condition (Range: 0-100)
36-Item Short-Form Health Survey | after 6weeks
  Qualify of life, The higher score means the better condition (Range: 0-100)
Geriatric Depression Scale | baseline
  Depression score, The higher score means the worse condition (Range: 0-15)
Geriatric Depression Scale | after 6weeks
  Depression score, The higher score means the worse condition (Range: 0-10)
Timed-Up and Go test | baseline
  Dynamic balance, The higher score means the worse balance.
Timed-Up and Go test | after 6weeks
  Dynamic balance, The higher score means the worse balance.
30s chair sit and stand | baseline
  Balance, The higher score means the better condition.
30s chair sit and stand | after 6weeks
  Balance, The higher score means the better condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided